Official Title of the Study: THE EFFECT OF VIDEO-ASSISTED ONLINE PREOPERATIVE EDUCATION ON FEAR, ANXIETY, SLEEP, AND STRESS IN PATIENTS UNDERGOING LAPAROSCOPIC CHOLECYSTECTOMY: A RANDOMIZED CONTROLLED TRIAL

**NCT Number:** Not Applicable (No NCT registration assigned)

**Document Date:** 16 June 2025

## **VOLUNTEER INFORMATION AND CONSENT FORM**

Dear Participant,

You have been invited to participate in a study titled "The Effect of Video-Assisted Online Preoperative Education on Fear, Anxiety, Sleep, and Stress in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Controlled Trial." Before deciding to participate, it is important for you to understand the purpose of the study, how it will be conducted, how your information will be used, and what the study entails. After you have been fully informed about the study and your questions have been answered, you will be asked to sign this form if you wish to participate

The purpose of this study was to examine the effects of online video-assisted video-assisted video-assisted video on fear, anxiety, sleep, and stress in patients undergoing gallbladder surgery during the preoperative period. Direct and objective markers of the surgical stress response were collected by blood samples to determine the effects on stress (serum cortisol) and blood sugar (serum glucose) levels. we aim.

The study participation criteria are; patients over 18 years of age, able to speak and write in Turkish, undergoing laparoscopic cholecystectomy for the first time, not receiving psychiatric treatment or taking medication, not having a chronic disease, not using cortisone-type medications, having a smartphone and knowing how to use it, having an anesthesia evaluation performed 1-3 days before surgery, and volunteering to participate in the study.

Once the decision to undergo surgery is made within the scope of the study, we will complete your consent form and assess your current state using fear, anxiety, sleep, and stress scales. After obtaining your consent, 3ml of blood will be drawn three times. Blood samples will be collected during your routine blood tests. These blood samples will be used to determine your stress level and blood sugar levels. No additional procedures will be performed for the blood draw. After receiving your contact information, we will video call you to provide information about the surgery, its techniques, the operating room environment, items you should have with you before your arrival, pre-operative bathing and grooming, the procedure for getting to the operating room, and answer your questions afterward. The total number of volunteers participating in the study is 128.

The expected benefits for you in this study are; to manage your fear, anxiety, sleep and stress before surgery, online video-supported training to reduce your physiological and psychological stress. It may also reduce postoperative recovery. This is not a risk anticipated for this study. There are no. Those whose surgery is canceled for any reason or those who withdraw from the study at any stage after volunteering to participate will not be included in the study. No specific medication/nutrient is prescribed for this study. It will not be recommended. If you wish to cancel the surgery due to complications, withdraw from the study at any stage after volunteering to participate in the study, You can stay.

To the research your participation for from you any One fee will not be wanted And accept the research you should in case of you One fee will not be paid. To the research Participation is voluntary. You will be given the right to withdraw after agreeing to participate in the study. The cost of the blood test to determine your stress hormone levels will not be charged to you or any official or private institution or organization under your protection. We plan to submit the study to TÜSEB as a TÜSEB project. No fees will be charged to patients for this research. If funding is

not provided, the costs of the research will be covered by the researcher. Participation in this research is entirely voluntary. You agree to participate in the research. You can refuse either in any One stage without research You can withdraw; even if you refuse or withdraw, your subsequent rights will be guaranteed. If you do not meet the inclusion criteria, you may be excluded from the study by the researcher, with your knowledge. In this case, your subsequent rights guarantee under will be taken. The research results scientific It will be used for the purpose; if you withdraw from the study or are removed by the researcher, your medical data may also be used for scientific purposes if necessary. All your medical and identity information will be kept confidential, and your identity will not be disclosed even if the study is published. However, research monitors, polling officers, ethics committees, and official authorities may access your medical information when necessary. You may also access your own medical information if you wish. You can reach.

If you encounter any problems during the research process, you can contact Nurse Instructor İzzettin EKİNCİ. Tel: 05424662246

Thank you for your participation and attention.

I HAVE READ THE ABOVE INFORMATION, AND HAVE BEEN GIVEN WRITTEN AND VERBAL EXPLANATIONS ABOUT THEM. UNDER THESE CONDITIONS, I AGREE TO PARTICIPATE IN THE RESEARCH WITH MY OWN CONSENT, WITHOUT ANY PRESSURE OR COERCION.

Volunteer's Name, Surname, Signature, Address (telephone number if available)

Name, Surname, Signature of the responsible researcher who conducted the research

# RESEARCH NAME: EFFECT OF VIDEO-ASSISTED ONLINE PREOPERATIVE EDUCATION ON FEAR, ANXIETY, SLEEP AND STRESS IN PATIENTS UNDERGOING LAPAROSCOPIC CHOLECYSTECTOMY: A RANDOMIZED CONTROLLED TRIAL

## **Dear Patient;**

We invite you to participate in a scientific study. As part of this scientific study, we will meet with you via phone/computer video call the night before your surgery. During this meeting, we will provide information about the surgery and assess your fear, anxiety, sleep, and stress levels. Additionally, when you arrive for anesthesia consent the day before your surgery, a nurse will draw your blood for routine blood tests from your arm, and we will also measure your stress hormone levels. After this blood draw, we will ask you a few questions. Whether you participate in the study will not affect your treatment or care in any way. You will not be charged for participation, and you will not be paid for the research. The results of this study will be published in scientific journals and discussed in scientific forums. Your information will not be disclosed anonymously in this study. Your information will be kept confidential and used solely for scientific purposes. You may not participate in this study at all; even if you do, you have the right to withdraw at any time at any stage. Participation in this study is entirely voluntary. If you volunteer to participate, you must answer the following survey questions. Answering the survey questions will take approximately 5-10 minutes. THANK YOU for your contributions to this scientific study.

#### INTRODUCTORY INFORMATION FORM

- 1. Date of birth (Specify the year.)
- a. Female b. Male
- 3. Marital status:
- a. Married b. Single
- 4. Your height? ..... cm
- **5. Your weight?** ..... kg
- 6. Educational status of the patient:
- a. Knows how to read and write b. Primary education c. Secondary education
- d. Associate degree e. Undergraduate f. Postgraduate
- 7. Working status:
- a. Working b. Not working c. Retired
- 8. Have you had any surgery before?
- a. Yes b. No

# PATIENT EVALUATION FORM (T0 EVALUATION)

**T0 Evaluation (Evaluation Made at the Anesthesia Approval Stage)** 

- 1. Serum Cortisol Level:
- 2. Serum Glucose Level:
- 3. Systolic Arterial Pressure:
- 4. Diastolic Arterial Pressure:
- 5. Pulse:
- 6. Respiratory rate:
- 7. SPO2:
- 8. Body temperature:
- 9. Surgical Fear Scale

This scale is designed to assess your fear of various aspects of a surgical procedure when you are about to undergo it. Please circle the option that best reflects how you currently feel.

# 1) I am afraid of surgery.

012345678910

I'm not afraid at all, I'm very afraid

# 2) I am afraid of anesthesia.

012345678910

I'm not afraid at all, I'm very afraid

# 3) I am afraid of post-operative pain.

012345678910

I'm not afraid at all, I'm very afraid

# 4) I am afraid of unpleasant side effects (such as nausea) after surgery.

012345678910

I'm not afraid at all, I'm very afraid

# 5) I am afraid that my health will deteriorate due to the surgery.

0 1 2 3 4 5 6 7 8 9 10

I'm not afraid at all, I'm very afraid

# 6) I am afraid that the surgery will be unsuccessful.

012345678910

I'm not afraid at all, I'm very afraid

# 7) I am afraid that I will not recover completely after the surgery.

0 1 2 3 4 5 6 7 8 9 10

I'm not afraid at all, I'm very afraid

# 8) I am afraid that my recovery process will be long after the surgery.

0 1 2 3 4 5 6 7 8 9 10

I'm not afraid at all, I'm very afraid

# 10. Visual Comparison Scale (VCS) Evaluation



# 11. RICHARD-CAMPBELL SLEEP SCALE

Below is a chart with scores ranging from 0 to 100 for each sleep statement. "0" represents the worst for each statement, and "100" represents the best. Please rate your perception of last night's sleep for each statement on the chart provided.

#### 1-My sleep last night

 $0--5--10--15--20--25--30--35--40--45--50--55--60--65--70--75--80--85--90--95--100 \\ It was light and deep$ 

#### 2-Falling asleep last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

I barely fell asleep I fell asleep almost as soon as I went to bed

#### 3- Frequency of waking up last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

I tossed and turned all night long, I didn't wake up much.

#### 4-Last night's awake time

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

Whenever I woke up or was woken up, I couldn't sleep. If I woke up, I fell asleep immediately.

#### 5-The quality of sleep last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

It was a bad night, I hardly slept at all. It was a good night, I never woke up.

## 6-Last night's noise level

**Total sleep perception Total Score of the Richard-Campbell Sleep Scale:** 

# PATIENT EVALUATION FORM (T1 EVALUATION)

T1 Assessment (Evaluation to be performed between 7:00-8:00 on the morning of surgery)

- 1. Serum Cortisol Level:
- 2. Serum Glucose Level:
- 3. Systolic Arterial Pressure:
- 4. Diastolic Arterial Pressure:
- 5. Pulse:
- 6. Respiratory rate:
- 7. SPO2:
- 8. Body temperature:
- 9. Surgical Fear Scale
- 10. Surgical Fear Scale

This scale is designed to assess your fear of various aspects of a surgical procedure when you are about to undergo it. Please circle the option that best reflects how you currently feel.

1) I am afraid of surgery.

012345678910

I'm not afraid at all, I'm very afraid

2) I am afraid of anesthesia.

012345678910

I'm not afraid at all, I'm very afraid

3) I am afraid of post-operative pain.

012345678910

I'm not afraid at all, I'm very afraid

4) I am afraid of unpleasant side effects (such as nausea) after surgery.

012345678910

I'm not afraid at all, I'm very afraid

5) I am afraid that my health will deteriorate due to the surgery.

0 1 2 3 4 5 6 7 8 9 10

I'm not afraid at all, I'm very afraid

6) I am afraid that the surgery will be unsuccessful.

012345678910

I'm not afraid at all, I'm very afraid

7) I am afraid that I will not recover completely after the surgery.

012345678910

I'm not afraid at all, I'm very afraid

8) I am afraid that my recovery process will be long after the surgery.

012345678910

I'm not afraid at all, I'm very afraid

11. Visual Comparison Scale (VCS) Evaluation



## 12. RICHARD-CAMPBELL SLEEP SCALE

Below is a chart with scores ranging from 0 to 100 for each sleep statement. "0" represents the worst for each statement, and "100" represents the best. Please rate your perception of last night's sleep for each statement on the chart provided.

## 1-My sleep last night

$$0--5--10--15--20--25--30--35--40--45--50--55--60--65--70--75--80--85--90--95--100$$
 It was light and deep

#### 2-Falling asleep last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

I barely fell asleep I fell asleep almost as soon as I went to bed

#### 3- Frequency of waking up last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

I tossed and turned all night long, I didn't wake up much.

#### 4-Last night's awake time

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

Whenever I woke up or was woken up, I couldn't sleep. If I woke up, I fell asleep immediately.

#### 5-The quality of sleep last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

It was a bad night, I hardly slept at all. It was a good night, I never woke up.

# 6-Last night's noise level

0---5---10---15---20---25---30---35---40---45---50---55---60---65---70---75---80---85---90---95---100 There was too much noise at night. There was too little noise at night.

**Total sleep perception Total Score of the Richard-Campbell Sleep Scale:** 

# PATIENT EVALUATION FORM (T 2 EVALUATION)

T2 Evaluation (Evaluation to be performed between 7:00-8:00 the day after surgery)

- 1. Serum Cortisol Level:
- 2. Serum Glucose Level:
- 3. Systolic Arterial Pressure:
- 4. Diastolic Arterial Pressure:
- 5. Pulse:
- 6. Respiratory rate:
- 7. SPO2:
- 8. Body temperature:
- 9. Surgical Fear Scale
- 10. Surgical Fear Scale

This scale is designed to assess your fear of various aspects of a surgical procedure when you are about to undergo it. Please circle the option that best reflects how you currently feel.

# 1) I am afraid of surgery.

0 1 2 3 4 5 6 7 8 9 10

I'm not afraid at all, I'm very afraid

# 2) I am afraid of anesthesia.

012345678910

I'm not afraid at all, I'm very afraid

# 3) I am afraid of post-operative pain.

012345678910

I'm not afraid at all, I'm very afraid

# 4) I am afraid of unpleasant side effects (such as nausea) after surgery.

012345678910

I'm not afraid at all, I'm very afraid

## 5) I am afraid that my health will deteriorate due to the surgery.

012345678910

I'm not afraid at all, I'm very afraid

# 6) I am afraid that the surgery will be unsuccessful.

 $0\ 1\ 2\ 3\ 4\ 5\ 6\ 7\ 8\ 9\ 10$ 

I'm not afraid at all, I'm very afraid

## 7) I am afraid that I will not recover completely after the surgery.

012345678910

I'm not afraid at all, I'm very afraid

## 8) I am afraid that my recovery process will be long after the surgery.

012345678910

I'm not afraid at all, I'm very afraid

# 11. Visual Comparison Scale (VCS) Evaluation



Hissedilebilecek En Viiksek Kavot

#### 12. RICHARD-CAMPBELL SLEEP SCALE

Below is a chart with scores ranging from 0 to 100 for each sleep statement. "0" represents the worst for each statement, and "100" represents the best. Please rate your perception of last night's sleep for each statement on the chart provided.

#### 1-My sleep last night

$$0--5--10--15--20--25--30--35--40--45--50--55--60--65--70--75--80--85--90--95--100$$
 It was light and deep

#### 2-Falling asleep last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

I barely fell asleep I fell asleep almost as soon as I went to bed

#### 3- Frequency of waking up last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

I tossed and turned all night long, I didn't wake up much.

## 4-Last night's awake time

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

Whenever I woke up or was woken up, I couldn't sleep. If I woke up, I fell asleep immediately.

#### 5-The quality of sleep last night

$$0 - -5 - -10 - -15 - -20 - -25 - -30 - -35 - -40 - -45 - -50 - -55 - -60 - -65 - -70 - -75 - -80 - -85 - -90 - -95 - -100$$

It was a bad night, I hardly slept at all. It was a good night, I never woke up.

#### 6-Last night's noise level

**Total sleep perception Total Score of the Richard-Campbell Sleep Scale:**